CLINICAL TRIAL: NCT00779792
Title: Comparison of Efficacy of Glycerol, Two Topical Steroids, and a Topical Immune Modulator Against Experimentally Induced Skin Irritation
Brief Title: Efficacy of Glycerol, Two Topical Steroids, and a Topical Immune Modulator Against Skin Irritation
Acronym: WA+TR_1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: LEO Pharma (Industry); University of Southern Denmark (Other)
Responsible Party: Anders Clemmensen, MD, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-001678-34
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-08

CONDITIONS: Dermatitis, Contact; Dermatitis, Occupational
Keywords: Irritant contact dermatitis; experimental contact dermatitis; treatment; efficacy; topical steroids; topical immune modulators; glycerol
MeSH Terms: conditions — Dermatitis, Contact; Dermatitis, Occupational; Dermatitis, Irritant | interventions — Clobetasol; Triamcinolone Acetonide; Tacrolimus; Glycerol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: clobetasol — 0.5 mg Clobetasol propionate (0.5 mg/g) ointment applied twice daily for 10 consecutive days
  Other Names: Dermovate
Drug: triamcinolone acetonide — 0.5 mg ointment twice daily for 10 consecutive days
  Other Names: Kenalog
Drug: tacrolimus — 0.5 mg tacrolimus ointment(0.1%) twice daily for 10 consecutive days
  Other Names: Protopic
Drug: glycerol — 0.5 mg glycerol ointment (20%) twice daily for 10 consecutive days
Drug: vehicle ointment (paraffin oil/soft white paraffin) — 0.5 mg vehicle ointment twice daily for 10 consecutive days

SUMMARY:
The purpose of this study is to compare the efficacy of glycerol ointment, triamcinolone acetonide ointment, clobetasol ointment and tacrolimus ointment on irritated skin in a cumulative skin irritation test model using healthy volunteers.

DETAILED DESCRIPTION:
Irritant contact dermatitis (ICD) is a frequent cause of hand eczema and occupational skin disease. One way to study ICD is to expose healthy volunteer skin to chemicals and evaluate the skin response. Because different chemicals act differently on the skin, the use of different skin irritants may provide more information than relying on one irritant only. In this study the two commonly used irritants sodium lauryl sulphate and nonanoic acid are exposed to the skin in a cumulative wash test. Treatment of ICD has classically involved topical steroids and/or emollients. However, the outcome is variable with some patients being very refractory to this regimen. This study was designed to investigate the relative efficacy of the steroids triamcinolone acetonide and clobetasol, the topical immune modulator tacrolimus, a 20% Glycerol ointment compared with an inert ointment vehicle on experimentally induced irritated skin.

ELIGIBILITY:
Inclusion Criteria:

* caucasian
* normal skin on both volar forearms
* oral and written informed consent

Exclusion Criteria:

* pregnant, lactating women
* no safe anticonceptive method used
* intake of systemic immunosuppressants (e.g. prednisolone)
* endocrine, immune, or liver disorders
* known allergy towards drugs applied to the skin

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
level of skin irritation as determined by visual reading, skin redness (color measurement), skin barrier integrity (transepidermal water loss measurement) and skin hydration (capacitance measurement) | End of treatment and summary measure (Area under the curve) of consecutive measurements at visit every other day for 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Anders Clemmensen, MD, Principal Investigator — Department of Dermatology, Odense University Hospital
Locations (1):
- Department of Dermatology, Odense University Hospital, Odense, Denmark

REFERENCES:
- [Background] Andersen F, Hedegaard K, Petersen TK, Bindslev-Jensen C, Fullerton A, Andersen KE. Comparison of the effect of glycerol and triamcinolone acetonide on cumulative skin irritation in a randomized trial. J Am Acad Dermatol. 2007 Feb;56(2):228-35. doi: 10.1016/j.jaad.2006.08.063. Epub 2006 Dec 6. PMID 17156893
- [Background] Schliemann S, Kelterer D, Bauer A, John SM, Skudlik C, Schindera I, Wehrmann W, Elsner P. Tacrolimus ointment in the treatment of occupationally induced chronic hand dermatitis. Contact Dermatitis. 2008 May;58(5):299-306. doi: 10.1111/j.1600-0536.2007.01314.x. PMID 18416762